CLINICAL TRIAL: NCT04825210
Title: Integrated Behavioral Health Prevention in Pediatric Primary Care for Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-1007
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Prevention
Keywords: Behavioral Health; Integrated Behavioral Health; Infant Self-Regulation; Parenting Skills

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Behavioral Health - Prevention (IBH-P) (Experimental): The IBH-P intervention addresses four areas: 1) assessment of emotional and behavioral adjustment, 2) parental education on important supports for emotional and behavioral health, 3) modeling and guidance on nurturing and responsive parenting, and 4) addressing parental concerns about and promoting child self-regulation. The primary focus of IBH-P is promoting infant self-regulation by teaching mothers how to soothe and calm their baby. Trauma-informed and relationship building methods are emphasized to acknowledge maternal experiences with violence and adversity and the desire to establish a strong working alliance. IBH-P is distinguished from Bright Futures through its emphasis on experiential learning, modeling of effective parenting skills, in-session practice and feedback, and proactive problem-solving. Families in IBH-P will receive all standard care elements of the well-child visit including pediatrician implementation of Bright Futures curriculum.
  Interventions: Behavioral: Integrated Behavioral Health - Prevention
- Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents, 4th Edition (Active Comparator): The Bright Futures control condition consists of standard of care in addressing emotional and behavioral health as provided by pediatricians. Pediatricians will follow the 4th edition of the Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents [pocket guide]. Guidelines are provided for topics to discuss and anticipatory guidance at each well-child visit. In contrast to IBH-P, there is an emphasis on didactic presentation, teaching mothers about developmental milestones, and responding to questions and concerns. These include discussions of crying, soothing, and feeding, although self-regulation is not a unifying theme.
  Interventions: Behavioral: Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents, 4th Edition

INTERVENTIONS:
Behavioral: Integrated Behavioral Health - Prevention — IBH-P consists of 15-30 minute visits with mothers as part of the 1, 2, 4, and 6 month well-child visits. The intervention is delivered by doctoral level pediatric psychologists that are an integrated member of the primary care team.
  Arms: Integrated Behavioral Health - Prevention (IBH-P)
Behavioral: Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents, 4th Edition — Bright Futures curriculum will be delivered by the pediatrician as part of the 1, 2, 4 and 6 month well-child visits.
  Arms: Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents, 4th Edition

SUMMARY:
The purpose of the study is to evaluate the acceptability and preliminary efficacy of a universal prevention program delivered by psychologists in conjunction with pediatric primary care well-child visits.

DETAILED DESCRIPTION:
Integrated behavioral health has emerged as an effective approach to addressing emotional and behavioral health needs of children in the pediatric setting, yet there is little evidence for a standardized model of care for providing universal preventive services in pediatric primary care. Current models are typically loosely constructed, inconsistently applied, and unspecified. Our aim is to evaluate a model of care developed to address these gaps. Integrated Behavioral Health-Prevention (IBH-P) is a collection of clinical strategies and structured approaches designed to promote emotional and behavioral health. IBH-P is delivered by psychologists in the pediatric setting as part of scheduled well-child visits. The overall objective of this study is to evaluate the efficacy of the intervention in promoting infant self-regulation. Maternal experience and satisfaction, adherence to well-child visits and immunizations will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Biological mother of a newborn infant presenting at the newborn well-child visit
* Intends to continue to receive infant's pediatric care at one of the three participating clinics over the next year.

Exclusion Criteria:

* Infant diagnosed as failure to thrive
* Infant exposure to illicit drugs in utero with the exception of THC
* Extensive care in the Neonatal Intensive Care Unit (>7 days)
* Child has other serious medical condition or acute psychosocial circumstances that results in child not receiving medical clearance from the pediatrician or psychologist for randomization
* mother or father of infant has received Building Futures intervention training

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Infant self-regulation | 7-month follow-up
  The Infant Behavior Questionnaire-Revised Very Short Form is a 36-item measure of three factors, positive affect, negative emotionality, and orienting/regulatory capacity. Scores range from 0 to 7, with higher scores representing greater positive affect, negative emotionality and orienting and regulatory capacity.
Parental knowledge of child development | 7-month follow-up
  The Knowledge of Infant Development Inventory is 58-item measure of caregiver knowledge of infant development. The total score will be calculated as the percentage of correct answers out of 58 items.
Maternal parenting behaviors | 7-month follow-up
  The Keys to Interactive Parenting Scale (KIPS) will be used to assess maternal parenting behaviors. KIPS is a structured observational measure and assesses 12 domains of parenting. The domains are scored on a 1 to 5-point scale with higher scores indicating higher quality parenting behaviors.

SECONDARY OUTCOMES:
Parenting beliefs and practices | 7-month follow-up
  The Baby Care Questionnaire is a 30-item measure of parenting belief and practices with 2 subscales, structure and attunement. Total scores range from 1 to 4 with higher scores indicating greater structure and attunement.
Maternal feelings of efficacy in infant care | 7-month follow-up
  The Maternal Self-Efficacy Scale is a 10-item self-report of feelings of efficacy in infant care. The total score will be used and ranges from 10 to 40 with higher scores representing greater maternal self-efficacy.
Maternal appraisement of life stress | 7-month follow-up
  The Perceived Stress Scale is a 14-item self-report of the degree to which situations in one's life within the past month are appraised as stressful. Scores range from 0 to 56 with higher scores indicating greater perceived stress.

OTHER OUTCOMES:
Maternal experiences of violence and adversity in childhood | Baseline
  The Philadelphia Urban Adverse Childhood Experiences is a 22-item self-report that will be used to measure maternal experience of childhood violence and adversity. The total score is a tally of the 22 items endorsed with higher scores indicating more experiences of violence and adversity.
Adherence to well-child visits in first 7 months of life | Infants' birth through 7-months of age
  The American Academy of Pediatrics recommends preventive pediatric care is provided across 5 visits in an infant's first 7 months of life. Percentage of adherence to the 5 well-child visits will be calculated.
Health Service Utilization - Immunizations | Infants' birth through 5-months of age
  Completion of immunizations at 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Ammerman, PhD, Principal Investigator — Cincinnati Children's Hospital Medical Center Cincinnati, OH USA
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the open science movement and with the directive of clinicaltrials.gov to include a data sharing plan in submissions, we will have the following data sharing policy: we will share with other investigators (1) all individual participant data after deidentification, and (2) study management documents (protocol, statistical analysis plan, consent form, analytic code, data dictionary).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and supporting information will be made available three months after publication of the primary article and ending five years after publication.
Access Criteria: Those requesting data will be required to submit a proposal to Robert.Ammerman@cchmc.org. This will be reviewed by the investigative team for methodological soundness and scientific merit before data is shared. This plan is consistent with guidelines developed by the International Committee of Medical Journal Editors (Taichman et al., 2017).

REFERENCES:
- [Background] Bright futures pocket guide (4th ed.). (2017). American Academy of Pediatrics.
- [Background] Putnam SP, Helbig AL, Gartstein MA, Rothbart MK, Leerkes E. Development and assessment of short and very short forms of the infant behavior questionnaire-revised. J Pers Assess. 2014;96(4):445-58. doi: 10.1080/00223891.2013.841171. Epub 2013 Nov 9. PMID 24206185
- [Background] MacPhee D. Knowledge of Infant Development Inventory: Manual. In. Colorado: Colorado State University; 2002.
- [Background] Winstanley A, Gattis M. The Baby Care Questionnaire: a measure of parenting principles and practices during infancy. Infant Behav Dev. 2013 Dec;36(4):762-75. doi: 10.1016/j.infbeh.2013.08.004. Epub 2013 Sep 18. PMID 24050932
- [Background] Teti DM, Gelfand DM. Behavioral competence among mothers of infants in the first year: the mediational role of maternal self-efficacy. Child Dev. 1991 Oct;62(5):918-29. doi: 10.1111/j.1467-8624.1991.tb01580.x. PMID 1756667
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Pachter LM, Lieberman L, Bloom SL, Fein JA. Developing a Community-Wide Initiative to Address Childhood Adversity and Toxic Stress: A Case Study of The Philadelphia ACE Task Force. Acad Pediatr. 2017 Sep-Oct;17(7S):S130-S135. doi: 10.1016/j.acap.2017.04.012. PMID 28865645
- [Background] Campo JV, Geist R, Kolko DJ. Integration of Pediatric Behavioral Health Services in Primary Care: Improving Access and Outcomes with Collaborative Care. Can J Psychiatry. 2018 Jul;63(7):432-438. doi: 10.1177/0706743717751668. Epub 2018 Apr 19. PMID 29673268
- [Background] Taichman DB, Sahni P, Pinborg A, Peiperl L, Laine C, James A, Hong ST, Haileamlak A, Gollogly L, Godlee F, Frizelle FA, Florenzano F, Drazen JM, Bauchner H, Baethge C, Backus J. Data Sharing Statements for Clinical Trials: A Requirement of the International Committee of Medical Journal Editors. Ann Intern Med. 2017 Jul 4;167(1):63-65. doi: 10.7326/M17-1028. Epub 2017 Jun 6. No abstract available. PMID 28586790